CLINICAL TRIAL: NCT04242680
Title: Improving Math Deficits in Children With Dyscalculia by tRNS: a Randomized, Double-blind Study
Brief Title: tRNS Combined to Cognitive Training in Children With Dyscalculia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Deny Menghini, Clinical Psychologist, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1547_OPBG_2018
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Developmental Dyscalculia
Keywords: Children; Adolescents; tRNS; transcranial random noise stimulation; EEG; numerical abilities; neurodevelopmental disorders; non-invasive brain stimulation; transcranial electrical stimulation
MeSH Terms: conditions — Dyscalculia; Neurodevelopmental Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brainstim DLPFC (Experimental): tRNS over bilateral DLPFC + cognitive training
  Interventions: Device: Brainstim DLPFC; Behavioral: Cognitive Training
- Brainstim PPC (Experimental): tRNS over bilateral PPC + cognitive training
  Interventions: Device: Brainstim PPC; Behavioral: Cognitive Training
- Brainstim Sham (Sham Comparator): Sham tRNS (bilateral DLPFC/bilateral PPC) + cognitive training
  Interventions: Device: Brainstim Sham; Behavioral: Cognitive Training

INTERVENTIONS:
Device: Brainstim DLPFC — The active tRNS will be delivered to bilateral DLPFC for five consecutive days for two weeks for a total of ten days.
  tRNS will be delivered by a battery driven, random-noise current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands.
  The electrodes will be placed on the left and right DLPFC, F3 and F4 position according to the 10-20 international EEG system for electrode placement, while participants will receive a usual treatment (cognitive training).
  Stimulation intensity will be set at 0.75 milliampere (mA) (100-500 Hz), the duration of stimulation will be 20 min.
  Other Names: tRNS over bilateral DLPFC
  Arms: Brainstim DLPFC
Device: Brainstim PPC — The active tRNS will be delivered to bilateral PPC for five consecutive days for two weeks for a total of ten days.
  tRNS will be delivered by a battery driven, random-noise current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands.
  The electrodes will be placed on the left and right PPC, P3 and P4 position according to the 10-20 international EEG system for electrode placement, while participants will receive a usual treatment (cognitive training).
  Stimulation intensity will be set at 0.75mA (100-500 Hz), the duration of stimulation will be 20 min.
  Other Names: tRNS over bilateral PPC
  Arms: Brainstim PPC
Device: Brainstim Sham — The same electrode placement will be used as in the stimulation conditions (Brainstim DLPFC or Brainstim PPC), but the current will be applied for 30 s and will be ramped down without the participants awareness, and will be held five consecutive days for two weeks for a total of ten days.
  Other Names: Sham tRNS (bilateral DLPFC/bilateral PPC)
  Arms: Brainstim Sham
Behavioral: Cognitive Training — A cognitive training (Vektor; Nemmi et al., 2016) will be adiministered concomitantly to Brainstim DLPFC, Brainstim PPC, Brainstim Sham for 20 min.
  The training consisted of math exercises (number line, calculations) and math-related exercises (visuo-spatial working memory, mental rotation).

SUMMARY:
The present study grounds on the absence of evidence-based treatment in individuals with developmental dyscalculia (DD). At this topic, the present study will explore the potential effect of transcranial random noise stimulation (tRNS) over dorsolateral prefrontal cortex (DLPFC) or posterior parietal cortex (PPC), cerebral areas usually disrupted in individuals with DD, in addition to a usual treatment such as cognitive training.

Therefore, the investigators hypothesized that active tRNS over DLPFC or PPC combined to cognitive training will boost math and math-related skills in children and adolescents with DD, modulating theta/beta ratio around stimulated cerebral network. On the contrary, sham tRNS (placebo) over DLPFC or PPC combined to cognitive training will not have significant effect in improving math skills. Further, both active and sham tRNS combined to cognitive training will be safe and well tolerated.

DETAILED DESCRIPTION:
The study design is randomized stratified, double blind, placebo-controlled.

A group of children and adolescents with DD will be selected and randomly assigned to three different conditions: 1. tRNS over bilateral DLPFC + cognitive training (Brainstim DLPFC); 2. tRNS over bilateral PPC (Brainstim PPC) + cognitive training; 3. sham tRNS (bilateral DLPFC/bilateral PPC; Brainstim Sham) + cognitive training.

In this project, the investigators will work to understand whether a brain-based intervention, with the use of tRNS, combined to a usual treatment can improve the outcome of individual with DD.

The protocol will allow the investigators to:

1. testing the critical role of two brain regions (DLPFC or PPC) usually involved in numerical abilities and disrupted in individuals with DD;
2. examining the neural changes (using EEG recordings) due to cognitive training without tRNS (Brainstim Sham) and with tRNS (Brainstim DLPFC; Brainstim PPC);
3. predicting training outcomes based on math-related skills;
4. testing the critical role of neural markers at developmental ages using a closed-loop tRNS to improve learning and cognitive outcomes from the training;
5. investigating the safety and tolerability of tRNS.

The investigator's overarching goal is to provide a scientific foundation for devising new rehabilitation strategies in DD.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with DD (Total Quotient of BDE-2 ≤ 70)
* IQ ≥ 85

Exclusion Criteria:

* Having a comorbidity with an important medical conditions;
* Having neurological diseases;
* Having Epilepsy o family history of epilepsy;
* Receiving a treatment for DD in the previous three months before the baseline screening;

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Number Line | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change of at least 1 SD in the "number line task" of the Diagnostic battery for Dyscalculia (BDE 2, Biancardi et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.

SECONDARY OUTCOMES:
Total Quotient | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the "Total Quotient" of the BDE 2 (Biancardi et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Numerical Quotient | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the "Numerical Quotient" of the BDE 2 (Biancardi et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Calculation Quotient | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the "Calculation Quotient" of the BDE 2 (Biancardi et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Number Sense Quotient | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the "Number Sense Quotient" of the BDE 2 (Biancardi et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Mental multiplications and additions | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the Mental Multiplications and Mental Additions tasks of the Diagnostic battery for Dyscalculia 1 (Biancardi et al., 2004) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Tempo Test Rekenen | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the total scores of the Tempo Test Rekenen (De Vos, 1992) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Geometric Puzzle | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the total scores of the Geometric Puzzle (Nepsy II, Korkman et al., 2011) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Math computerized task | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in a math computerized task (Math Proc, PEBL) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Motivation and study strategies Questionnaire | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change (lower score means better outcome) in the Motivation and study strategies Questionnaire from 8 to 15 ages (AMOS 8-15, Cornoldi et al., 2005) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Math Anxiety Questionnaire | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change (lower score means better outcome) in the Math Anxiety Questionnaire (MARS, Saccani and Cornoldi, 2005) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Sleep quality | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change (lower score means better outcome) in the Sleep Disturbance Scale for Children (SDSC, Bruni et al., 1996) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Parental stress | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change (higher score means better outcome) in the Parent Stress Index (PSI, Guarino et al., 2014) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Emotional/behavioural problems | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change (lower score means better outcome) in the Cross-symptom assessment scales of the Kiddie-Sads- present and lifetime version-Diagnostic and Statistical Manual of Mental Disorders 5 (K-SADS- DSM-5, Kaufman et al., 2016) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Math improvement at school | three months after the intervention
  The proportion of patients with change in math markers in the transcript (scale from 0 to 10, where 10 is the best level and 0 the worst) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Theta/Beta ratio | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with reduction of theta/beta ratio in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Verbal and visuo-spatial working-memory | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the index of verbal and visuo-spatial n-back (more score means better outcome) in Brainstim DLPFC and Brainstim PPC than in Brainstim Sham.
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | immediately after the intervention, one week and three months after the intervention
  The proportion of patients with change in the questionnaire of safety and tolerability (Questionnaire of adverse effect; Brunoni et al., 2011) in Brainstim DLPFC and Brainstim PPC will be the same than in Brainstim Sham.

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital and Research Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APA (2013). Diagnostic and statistical manual of mental disorders: DSM 5. Washington, DC: American Psychiatric Association.
- [Background] Baroody, AJ., Tiilikainen, SH. Two perspectives on addition development. In: Baroody AJ, Dowker A, editors. The development of arithmetic concepts and skills: The construction of adaptive expertise. Erlbaum; Mahwah, NJ: 2003. pp. 75-125.
- [Background] Belacchi, C., Scalisi, T.G., Cannoni, E. e Cornoldi, C. (2008). Matrici Progressive di Raven Forma
- [Background] Biancardi, A., Bachmann, C., Nicoletti, C. (2016) BDE 2 - Batteria discalculia evolutiva Test per la diagnosi dei disturbi dell'elaborazione numerica e del calcolo in età evolutiva - 8-13 anni.
- [Background] Cornoldi, C., Colpo, G. (2012). Prove di Lettura MT per la Scuola Elementare-2, Firenze, Organizzazioni Speciali.
- [Background] Lehto, J.E. et al. (2003). Dimensions of executive functioning: Evidence from children. British Journal of Developmental Psychology, 21, 59-80.
- [Background] Sartori, G., Job, R., Tressoldi, PE. (2007). DDE-2. Batteria per la valutazione della dislessia e della disortografia evolutiva, Firenze, Organizzazioni Speciali.
- [Result] Ambrus GG, Paulus W, Antal A. Cutaneous perception thresholds of electrical stimulation methods: comparison of tDCS and tRNS. Clin Neurophysiol. 2010 Nov;121(11):1908-14. doi: 10.1016/j.clinph.2010.04.020. Epub 2010 May 14. PMID 20471313
- [Result] Ansari D. Effects of development and enculturation on number representation in the brain. Nat Rev Neurosci. 2008 Apr;9(4):278-91. doi: 10.1038/nrn2334. PMID 18334999
- [Result] Arsalidou M, Taylor MJ. Is 2+2=4? Meta-analyses of brain areas needed for numbers and calculations. Neuroimage. 2011 Feb 1;54(3):2382-93. doi: 10.1016/j.neuroimage.2010.10.009. Epub 2010 Oct 12. PMID 20946958
- [Result] Butterworth B. Foundational numerical capacities and the origins of dyscalculia. Trends Cogn Sci. 2010 Dec;14(12):534-41. doi: 10.1016/j.tics.2010.09.007. PMID 20971676
- [Result] Butterworth B, Varma S, Laurillard D. Dyscalculia: from brain to education. Science. 2011 May 27;332(6033):1049-53. doi: 10.1126/science.1201536. PMID 21617068
- [Result] Cantlon JF, Brannon EM, Carter EJ, Pelphrey KA. Functional imaging of numerical processing in adults and 4-y-old children. PLoS Biol. 2006 May;4(5):e125. doi: 10.1371/journal.pbio.0040125. Epub 2006 Apr 11. PMID 16594732
- [Result] Cappelletti M, Gessaroli E, Hithersay R, Mitolo M, Didino D, Kanai R, Cohen Kadosh R, Walsh V. Transfer of cognitive training across magnitude dimensions achieved with concurrent brain stimulation of the parietal lobe. J Neurosci. 2013 Sep 11;33(37):14899-907. doi: 10.1523/JNEUROSCI.1692-13.2013. PMID 24027289
- [Result] Chaieb L, Antal A, Pisoni A, Saiote C, Opitz A, Ambrus GG, Focke N, Paulus W. Safety of 5 kHz tACS. Brain Stimul. 2014 Jan-Feb;7(1):92-6. doi: 10.1016/j.brs.2013.08.004. Epub 2013 Sep 13. PMID 24064065
- [Result] Cohen Kadosh R, Cohen Kadosh K, Schuhmann T, Kaas A, Goebel R, Henik A, Sack AT. Virtual dyscalculia induced by parietal-lobe TMS impairs automatic magnitude processing. Curr Biol. 2007 Apr 17;17(8):689-93. doi: 10.1016/j.cub.2007.02.056. Epub 2007 Mar 22. PMID 17379521
- [Result] Cohen Kadosh R, Lammertyn J, Izard V. Are numbers special? An overview of chronometric, neuroimaging, developmental and comparative studies of magnitude representation. Prog Neurobiol. 2008 Feb;84(2):132-47. doi: 10.1016/j.pneurobio.2007.11.001. Epub 2007 Nov 19. PMID 18155348
- [Result] Collins A, Koechlin E. Reasoning, learning, and creativity: frontal lobe function and human decision-making. PLoS Biol. 2012;10(3):e1001293. doi: 10.1371/journal.pbio.1001293. Epub 2012 Mar 27. PMID 22479152
- [Result] Costanzo F, Menghini D, Caltagirone C, Oliveri M, Vicari S. High frequency rTMS over the left parietal lobule increases non-word reading accuracy. Neuropsychologia. 2012 Sep;50(11):2645-51. doi: 10.1016/j.neuropsychologia.2012.07.017. Epub 2012 Jul 20. PMID 22820638
- [Result] Costanzo F, Menghini D, Caltagirone C, Oliveri M, Vicari S. How to improve reading skills in dyslexics: the effect of high frequency rTMS. Neuropsychologia. 2013 Dec;51(14):2953-9. doi: 10.1016/j.neuropsychologia.2013.10.018. Epub 2013 Oct 31. PMID 24184439
- [Result] Costanzo F, Rossi S, Varuzza C, Varvara P, Vicari S, Menghini D. Long-lasting improvement following tDCS treatment combined with a training for reading in children and adolescents with dyslexia. Neuropsychologia. 2019 Jul;130:38-43. doi: 10.1016/j.neuropsychologia.2018.03.016. Epub 2018 Mar 14. PMID 29550525
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Giacomo K, Vicari S, Menghini D. Evidence for reading improvement following tDCS treatment in children and adolescents with Dyslexia. Restor Neurol Neurosci. 2016;34(2):215-26. doi: 10.3233/RNN-150561. PMID 26890096
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Koch G, Vicari S, Menghini D. Reading changes in children and adolescents with dyslexia after transcranial direct current stimulation. Neuroreport. 2016 Mar 23;27(5):295-300. doi: 10.1097/WNR.0000000000000536. PMID 26848997
- [Result] Dehaene S. Origins of mathematical intuitions: the case of arithmetic. Ann N Y Acad Sci. 2009 Mar;1156:232-59. doi: 10.1111/j.1749-6632.2009.04469.x. PMID 19338511
- [Result] Dehaene S, Spelke E, Pinel P, Stanescu R, Tsivkin S. Sources of mathematical thinking: behavioral and brain-imaging evidence. Science. 1999 May 7;284(5416):970-4. doi: 10.1126/science.284.5416.970. PMID 10320379
- [Result] Delazer M, Domahs F, Bartha L, Brenneis C, Lochy A, Trieb T, Benke T. Learning complex arithmetic--an fMRI study. Brain Res Cogn Brain Res. 2003 Dec;18(1):76-88. doi: 10.1016/j.cogbrainres.2003.09.005. PMID 14659499
- [Result] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Result] Fertonani A, Pirulli C, Miniussi C. Random noise stimulation improves neuroplasticity in perceptual learning. J Neurosci. 2011 Oct 26;31(43):15416-23. doi: 10.1523/JNEUROSCI.2002-11.2011. PMID 22031888
- [Result] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Result] Hauser TU, Rotzer S, Grabner RH, Merillat S, Jancke L. Enhancing performance in numerical magnitude processing and mental arithmetic using transcranial Direct Current Stimulation (tDCS). Front Hum Neurosci. 2013 Jun 6;7:244. doi: 10.3389/fnhum.2013.00244. eCollection 2013. PMID 23761750
- [Result] Heth I, Lavidor M. Improved reading measures in adults with dyslexia following transcranial direct current stimulation treatment. Neuropsychologia. 2015 Apr;70:107-13. doi: 10.1016/j.neuropsychologia.2015.02.022. Epub 2015 Feb 19. PMID 25701796
- [Result] Hyde DC, Boas DA, Blair C, Carey S. Near-infrared spectroscopy shows right parietal specialization for number in pre-verbal infants. Neuroimage. 2010 Nov 1;53(2):647-52. doi: 10.1016/j.neuroimage.2010.06.030. Epub 2010 Jun 16. PMID 20561591
- [Result] Isaacs EB, Edmonds CJ, Lucas A, Gadian DG. Calculation difficulties in children of very low birthweight: a neural correlate. Brain. 2001 Sep;124(Pt 9):1701-7. doi: 10.1093/brain/124.9.1701. PMID 11522573
- [Result] Iuculano T, Cohen Kadosh R. Preliminary evidence for performance enhancement following parietal lobe stimulation in Developmental Dyscalculia. Front Hum Neurosci. 2014 Feb 7;8:38. doi: 10.3389/fnhum.2014.00038. eCollection 2014. PMID 24570659
- [Result] Kaufmann L, Mazzocco MM, Dowker A, von Aster M, Gobel SM, Grabner RH, Henik A, Jordan NC, Karmiloff-Smith AD, Kucian K, Rubinsten O, Szucs D, Shalev R, Nuerk HC. Dyscalculia from a developmental and differential perspective. Front Psychol. 2013 Aug 21;4:516. doi: 10.3389/fpsyg.2013.00516. eCollection 2013. No abstract available. PMID 23970870
- [Result] Kaufmann L, Wood G, Rubinsten O, Henik A. Meta-analyses of developmental fMRI studies investigating typical and atypical trajectories of number processing and calculation. Dev Neuropsychol. 2011;36(6):763-87. doi: 10.1080/87565641.2010.549884. PMID 21761997
- [Result] Korkman, M., Kirk, U., Kemp, S. (2011). NEPSY-II. Giunti, OS.
- [Result] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Result] Kucian K, Loenneker T, Dietrich T, Dosch M, Martin E, von Aster M. Impaired neural networks for approximate calculation in dyscalculic children: a functional MRI study. Behav Brain Funct. 2006 Sep 5;2:31. doi: 10.1186/1744-9081-2-31. PMID 16953876
- [Result] Looi CY, Duta M, Brem AK, Huber S, Nuerk HC, Cohen Kadosh R. Combining brain stimulation and video game to promote long-term transfer of learning and cognitive enhancement. Sci Rep. 2016 Feb 23;6:22003. doi: 10.1038/srep22003. PMID 26902664
- [Result] Looi CY, Lim J, Sella F, Lolliot S, Duta M, Avramenko AA, Cohen Kadosh R. Transcranial random noise stimulation and cognitive training to improve learning and cognition of the atypically developing brain: A pilot study. Sci Rep. 2017 Jul 5;7(1):4633. doi: 10.1038/s41598-017-04649-x. PMID 28680099
- [Result] Mattai A, Miller R, Weisinger B, Greenstein D, Bakalar J, Tossell J, David C, Wassermann EM, Rapoport J, Gogtay N. Tolerability of transcranial direct current stimulation in childhood-onset schizophrenia. Brain Stimul. 2011 Oct;4(4):275-80. doi: 10.1016/j.brs.2011.01.001. Epub 2011 Feb 1. PMID 22032743
- [Result] Miniussi C, Rossini PM. Transcranial magnetic stimulation in cognitive rehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):579-601. doi: 10.1080/09602011.2011.562689. Epub 2011 Jun 24. PMID 21462081
- [Result] Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD. The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cogn Psychol. 2000 Aug;41(1):49-100. doi: 10.1006/cogp.1999.0734. PMID 10945922
- [Result] Pasqualotto A. Transcranial random noise stimulation benefits arithmetic skills. Neurobiol Learn Mem. 2016 Sep;133:7-12. doi: 10.1016/j.nlm.2016.05.004. Epub 2016 May 17. PMID 27224886
- [Result] Popescu T, Krause B, Terhune DB, Twose O, Page T, Humphreys G, Cohen Kadosh R. Transcranial random noise stimulation mitigates increased difficulty in an arithmetic learning task. Neuropsychologia. 2016 Jan 29;81:255-264. doi: 10.1016/j.neuropsychologia.2015.12.028. Epub 2015 Dec 28. PMID 26731199
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Price GR, Holloway I, Rasanen P, Vesterinen M, Ansari D. Impaired parietal magnitude processing in developmental dyscalculia. Curr Biol. 2007 Dec 18;17(24):R1042-3. doi: 10.1016/j.cub.2007.10.013. PMID 18088583
- [Result] Rivera SM, Reiss AL, Eckert MA, Menon V. Developmental changes in mental arithmetic: evidence for increased functional specialization in the left inferior parietal cortex. Cereb Cortex. 2005 Nov;15(11):1779-90. doi: 10.1093/cercor/bhi055. Epub 2005 Feb 16. PMID 15716474
- [Result] Rotzer S, Kucian K, Martin E, von Aster M, Klaver P, Loenneker T. Optimized voxel-based morphometry in children with developmental dyscalculia. Neuroimage. 2008 Jan 1;39(1):417-22. doi: 10.1016/j.neuroimage.2007.08.045. Epub 2007 Sep 7. PMID 17928237
- [Result] Rubio-Morell B, Rotenberg A, Hernandez-Exposito S, Pascual-Leone A. [The use of noninvasive brain stimulation in childhood psychiatric disorders: new diagnostic and therapeutic opportunities and challenges]. Rev Neurol. 2011 Aug 16;53(4):209-25. Spanish. PMID 21780073
- [Result] Snowball A, Tachtsidis I, Popescu T, Thompson J, Delazer M, Zamarian L, Zhu T, Cohen Kadosh R. Long-term enhancement of brain function and cognition using cognitive training and brain stimulation. Curr Biol. 2013 Jun 3;23(11):987-92. doi: 10.1016/j.cub.2013.04.045. Epub 2013 May 16. PMID 23684971
- [Result] Stanescu-Cosson R, Pinel P, van De Moortele PF, Le Bihan D, Cohen L, Dehaene S. Understanding dissociations in dyscalculia: a brain imaging study of the impact of number size on the cerebral networks for exact and approximate calculation. Brain. 2000 Nov;123 ( Pt 11):2240-55. doi: 10.1093/brain/123.11.2240. PMID 11050024
- [Result] Terney D, Chaieb L, Moliadze V, Antal A, Paulus W. Increasing human brain excitability by transcranial high-frequency random noise stimulation. J Neurosci. 2008 Dec 24;28(52):14147-55. doi: 10.1523/JNEUROSCI.4248-08.2008. PMID 19109497
- [Result] Turkeltaub PE, Benson J, Hamilton RH, Datta A, Bikson M, Coslett HB. Left lateralizing transcranial direct current stimulation improves reading efficiency. Brain Stimul. 2012 Jul;5(3):201-207. doi: 10.1016/j.brs.2011.04.002. Epub 2011 May 5. PMID 22305346